CLINICAL TRIAL: NCT00472940
Title: Prevalence of Hypogonadism in Male Cancer Patients
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Marco Marcelli, Professor, Medicine-Endocrinology, Baylor College of Medicine
Other Study IDs: H-19709
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Cancer; Hypogonadism
Keywords: Cancer; Hypogonadism; testosterone; cachexia
MeSH Terms: conditions — Neoplasms; Hypogonadism; Cachexia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cancer and its complications are common problems. In most cases, this condition has a profound impact on survival and quality of life (QoL). Fatigue, sexual dysfunction, decreased sexual drive, depression and poor appetite are commonly seen in these patients. However, these symptoms also are seen in men with other conditions including those with low testosterone levels.

The objective of this study is to determine the number of male patients with cancer that have low testosterone levels and to establish the relationship between testosterone levels and the symptoms that these patients experience.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥ 18 years of age with histological diagnosis of cancer for cancer group.
2. Provide written informed consent prior to screening.
3. Histological diagnosis of cancer other than non-melanoma skin cancer for the two cancer groups.

Exclusion Criteria:

1. Concomitant use of GH, Megestrol, Marinol, or any other anabolic agent, appetite stimulant (including corticosteroids other than dexamethasone at the time of IV chemotherapy administrations), tube feedings, or parenteral nutrition during the 3 months prior to entering the study.
2. Participation in a clinical trial with investigational agents within 1 month of enrollment.
3. Prior or current use of other medications that interfere with gonadal axis (androgens, estrogens, anti-androgens, etc).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male subjects with cancer and non-cancer controls
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2006-11; Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Garcia, MD, Principal Investigator — Baylor College of Medicine, Michael E. DeBakey VAMC
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Garcia JM, Li H, Mann D, Epner D, Hayes TG, Marcelli M, Cunningham GR. Hypogonadism in male patients with cancer. Cancer. 2006 Jun 15;106(12):2583-91. doi: 10.1002/cncr.21889. PMID 16688773
- [Derived] Burney BO, Hayes TG, Smiechowska J, Cardwell G, Papusha V, Bhargava P, Konda B, Auchus RJ, Garcia JM. Low testosterone levels and increased inflammatory markers in patients with cancer and relationship with cachexia. J Clin Endocrinol Metab. 2012 May;97(5):E700-9. doi: 10.1210/jc.2011-2387. Epub 2012 Mar 14. PMID 22419719